CLINICAL TRIAL: NCT06661187
Title: The Effect of Using Simple Psychological Interventions and Cryoanalgesia for Reducing Arterial Puncture Pain and Anxiety in Critically Ill Patients
Brief Title: Simple Psychological Interventions and Cryoanalgesia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Cryoanalgesia
Record Dates: First submitted 2024-10-19; First posted 2024-10-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-10

CONDITIONS: Arterial Puncture
Keywords: Cryoanalgesia; Arterial Puncture; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: group one will use cryoanalgesia group two will use simple psychological instruction control group Group will use both method (cryoanalgesia and simple psychological instruction)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cryoanalgesia (Experimental): Patients who received cryoanalgesia: patients subjects underwent arterial puncture. patients in the intervention group had a small plastic bag filled with 12 oz of crushed ice applied to the radial artery puncture site for 3 min (timed with a stopwatch) without external compression or massage.
  Interventions: Procedure: Cryoanalgesia
- Psychological instructions (Experimental): Psychological interventions using verbal signals of the impending procedure, music distraction, visual distraction, and breathing interventions be used during arterial puncture injections in adults
  Interventions: Procedure: Psychological instructions
- control group (Placebo Comparator): Patients received routine care
  Interventions: Procedure: Routine care
- Mixed group (Active Comparator): received both interventions
  Interventions: Procedure: Cryoanalgesia; Procedure: Psychological instructions

INTERVENTIONS:
Procedure: Cryoanalgesia — Patients who received cryoanalgesia: patients subjects underwent arterial puncture. patients in the intervention group had a small plastic bag filled with 12 oz of crushed ice applied to the radial artery puncture site for 3 min (timed with a stopwatch) without external compression or massage.
  Arms: Cryoanalgesia; Mixed group
Procedure: Psychological instructions — Psychological interventions using verbal signals of the impending procedure, music distraction, visual distraction, and breathing interventions be used during arterial puncture in adults
  Arms: Mixed group; Psychological instructions
Procedure: Routine care — No intervention deliver routine care
  Arms: control group

SUMMARY:
This study aims to explore the effect of using simple psychological interventions and cryoanalgesia for reducing arterial punctures pain and anxiety in critically ill patients

DETAILED DESCRIPTION:
The present study will be carried out in two interventions Patients who received cryoanalgesia: patients subjects underwent arterial puncture. patients in the intervention group had a small plastic bag filled with 12 oz of crushed ice applied to the radial artery puncture site for 3 min (timed with a stopwatch) without external compression or massage.

Psychological interventions using verbal signals of the impending procedure, music distraction, visual distraction, and breathing interventions be used during arterial puncture in adults

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both genders.
* Consciousness patient required arterial puncture

Exclusion Criteria:

* Unconsciousness patients Patients with complicated site from arterial puncture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Severity of pain using numerical pain scale | Three observations after the end arterial puncture procedure
  The patient is asked to rate their pain on a 0-10 scale, where: 0 = No pain 1-3 = Mild pain (nagging, annoying, but doesn't interfere much with daily activities) 4-6 = Moderate pain (noticeable, bothersome, may interfere with concentration or some activities) 7-10 = Severe pain (very intense, disabling, interferes with most activities or rest)
Level of anxiety using the Hamilton Anxiety Rating Scale | Two observations before and after arterial puncture procedure
  Hamilton Anxiety Rating Scale consisted of 14 items measuring psychic anxiety (mental agitation) and somatic anxiety (physical complaints) Each item scored from 0 (not present) to 4 (severe) Total score ranges from 0-56, with higher scores indicating more severe

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Damanhour university, Damanhūr
  - Faculty Of Nursing, Damanhūr